CLINICAL TRIAL: NCT05088161
Title: Prognostic Biomarkers of Pancreatic Cancer Based on Proteomics Techniques
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: JJDB-SR-2021-02
Record Dates: First submitted 2021-06-23; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we will use high-throughput proteomics techniques to search for biomarkers of post-operative prognosis of pancreatic cancer in samples of patients who have been diagnosed with pancreatic cancer through bioinformatics analysis.

DETAILED DESCRIPTION:
This study plan from the affiliated hospital of Qingdao university collected 20 cases of patients with pancreatic cancer pathological tissue samples and clinical data, including clinical diagnostic information, laboratory tests, imaging examination results and other information data), through high-throughput proteomic technology in pancreatic cancer pathological finding biomarkers, the bioinformatics analysis to explore the prognosis biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Chinese nationality, age and gender are not limited.
* Pathologically confirmed pancreatic cancer patients.
* Pathological specimens were archived tumor tissue samples after a diagnosis of pancreatic cancer.
* Clinical diagnostic information was complete three months before sampling.

Exclusion Criteria:

* Patients with a second primary tumor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects in this study were all patients with pathologically diagnosed pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-11-12 (Estimated); Study Completion 2022-03-12 (Estimated)

PRIMARY OUTCOMES:
Differentially expressed proteins in tumor and paracancer tissues | 180 Days
  Two dimensional gel electrophoresis, mass spectrometry and other techniques were used to separate and compare pancreatic cancer tissues and normal adjacent tissues to search for differentially expressed proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No